CLINICAL TRIAL: NCT00154310
Title: Multi-center, Open-label, Prospective, Randomized, Parallel Group Study Investigating a CNI-free Regimen With Enteric-Coated Mycophenolate Sodium (EC-MPS) and Everolimus in Comparison to Standard Therapy With Enteric-Coated Mycophenolate Sodium (EC-MPS) and Cyclosporine Microemulsion in de Novo Renal Transplant Patients
Brief Title: Efficacy and Safety of Everolimus With Enteric-Coated Mycophenolate Sodium (EC-MPS) in a Cyclosporine Microemulsion-free Regimen Compared to Standard Therapy in de Novo Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001A2418
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-10

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, everolimus, immunosuppressants, CNI-free
MeSH Terms: interventions — Everolimus; Cyclosporine; Mycophenolic Acid; Adrenal Cortex Hormones

ARMS (2):
- Everolimus + Mycophenolate sodium (Experimental): Everolimus tablets orally twice a day to maintain a level of 6- 10 ng/mL and enteric-coated mycophenolate sodium orally twice a day to achieve a target dose of 1440 mg/day. Corticosteroids were added to the immunosuppressive regimen with a minimum dose of 5 mg prednisolone or equivalent and had to be continued throughout the first year. Cyclosporine withdrawal started from Month 4.5 post-transplant.
  Interventions: Drug: Everolimus; Drug: Enteric-coated mycophenolate sodium; Drug: Corticosteroids
- Cyclosporine + Mycophenolate sodium (Active Comparator): Cyclosporine tablets orally twice a day to achieve protocol specific target levels and enteric-coated mycophenolate sodium orally twice a day to achieve a target dose of 1440 mg/day. Corticosteroids were added to the immunosuppressive regimen with a minimum dose of 5mg prednisolone or equivalent and had to be continued throughout the first year.
  Interventions: Drug: Cyclosporine; Drug: Enteric-coated mycophenolate sodium; Drug: Corticosteroids

INTERVENTIONS:
Drug: Everolimus — Everolimus tablets orally twice a day to maintain a level of 6- 10 ng/mL.
  Other Names: certican
  Arms: Everolimus + Mycophenolate sodium
Drug: Cyclosporine — Tablets orally twice a day to maintain protocol specific target blood levels
  Other Names: Sandimmun Optoral
  Arms: Cyclosporine + Mycophenolate sodium
Drug: Enteric-coated mycophenolate sodium — Enteric-coated mycophenolate sodium orally twice a day to achieve a target dose of 1440 mg/day.
  Other Names: Myfortic
Drug: Corticosteroids — Corticosteroids were added to the immunosuppressive regimen with a minimum dose of 5mg prednisolone or equivalent and had to be continued throughout the first year.

SUMMARY:
The purpose of this study is to assess whether a calcineurin inhibitor (CNI)-free regimen with enteric-coated mycophenolate sodium (EC-MPS) and everolimus is as safe and well-tolerated as the standard regimen containing enteric-coated mycophenolate sodium (EC-MPS) and cyclosporine microemulsion, but results in better renal function.

ELIGIBILITY:
Inclusion Criteria :

The following inclusion criteria had to be present at BL 1 (Screening visit prior to transplantation):

1. Males or females, aged 18 - 65 years
2. Recipients of de novo cadaveric, living unrelated or living related kidney transplants
3. Females capable of becoming pregnant must have a negative serum pregnancy test within 7 days prior to or at BL 1, and are required to practice an approved method of birth control for the duration of the study and for a period of 6 weeks following discontinuation of study medication, even where there has been a history of infertility
4. Patients who are willing and able to participate in the study and from whom written informed consent has been obtained

   Of all patients included into the study at BL 1 (prior to transplantation), those who continued into the randomized study period had to meet the following condition at BL 2, prior to randomization:
5. Patients had to be on an immunosuppressive regimen with EC-MPS (target dose; 1440 mg/day, if tolerated; minimal dose: 720 mg/day), cyclosporine and corticosteroids
6. Patients with an actual serum creatinine =< 3.0 mg/dl

Exclusion Criteria:

The following exclusion criteria must not be present at BL 1 (Screening visit prior to transplantation):

1. More than one previous renal transplantation
2. Multi-organ recipients (e.g., kidney and pancreas) or previous transplant with any other organ, different from kidney
3. Graft loss due to immunological reasons in the first year after transplantation (in case of secondary transplantation)
4. Patients who are recipients of A-B-O incompatible transplants
5. Patients with a historical or current peak PRA of > 25%
6. Patients with already existing antibodies against the HLA-type of the receiving transplant
7. Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception

   Of all patients included into the study at BL 1 (prior to transplantation), those who met one or more of the following criteria at BL 2, prior to randomization, should not continue into the randomized study period:
8. Graft loss or death
9. Changes to the immunosuppressive regimen prior to randomization due to immunologic reasons
10. Patients who suffered from severe rejection (>= BANFF II acute rejection), recurrent acute rejection, or steroid resistant acute rejection
11. Proteinuria > 1g/day

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (3):
- Novartis Investigational Sites, Nuremberg, Germany
- Switzerland (2):
  - Novartis Pharma AG, Basel
  - Novartis Investigational Sites, Bern

REFERENCES:
- [Derived] Sommerer C, Witzke O, Lehner F, Arns W, Reinke P, Eisenberger U, Vogt B, Heller K, Jacobi J, Guba M, Stahl R, Hauser IA, Kliem V, Wuthrich RP, Muhlfeld A, Suwelack B, Duerr M, Paulus EM, Zeier M, Porstner M, Budde K; ZEUS and HERAKLES study investigators. Onset and progression of diabetes in kidney transplant patients receiving everolimus or cyclosporine therapy: an analysis of two randomized, multicenter trials. BMC Nephrol. 2018 Sep 19;19(1):237. doi: 10.1186/s12882-018-1031-1. PMID 30231851
- [Derived] Eisenberger U, Budde K, Lehner F, Sommerer C, Reinke P, Witzke O, Wuthrich RP, Stahl R, Heller K, Suwelack B, Muhlfeld A, Hauser IA, Nadalin S, Porstner M, Arns W; ZEUS Study Investigators. Histological findings to five years after early conversion of kidney transplant patients from cyclosporine to everolimus: an analysis from the randomized ZEUS study. BMC Nephrol. 2018 Jun 28;19(1):154. doi: 10.1186/s12882-018-0950-1. PMID 29954336
- [Derived] Lehner F, Budde K, Zeier M, Wuthrich RP, Reinke P, Eisenberger U, Muhlfeld A, Arns W, Stahl R, Heller K, Witzke O, Wolters HH, Suwelack B, Klehr HU, Stangl M, Hauser IA, Nadalin S, Porstner M, May C, Paulus EM, Sommerer C; ZEUS Study Investigators. Efficacy and safety of conversion from cyclosporine to everolimus in living-donor kidney transplant recipients: an analysis from the ZEUS study. Transpl Int. 2014 Nov;27(11):1192-204. doi: 10.1111/tri.12411. Epub 2014 Aug 20. PMID 25070687
- [Derived] Budde K, Becker T, Arns W, Sommerer C, Reinke P, Eisenberger U, Kramer S, Fischer W, Gschaidmeier H, Pietruck F; ZEUS Study Investigators. Everolimus-based, calcineurin-inhibitor-free regimen in recipients of de-novo kidney transplants: an open-label, randomised, controlled trial. Lancet. 2011 Mar 5;377(9768):837-47. doi: 10.1016/S0140-6736(10)62318-5. Epub 2011 Feb 19. PMID 21334736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an open-label, randomized, parallel-group, multi-center study with two treatment groups, cyclosporine continuation and cyclosporine withdrawal starting from Month 4.5 post-transplant. Study started in June 2005 and ended in September 2008.
Period: Overall Study
Arm/Group | Everolimus + Mycophenolate Sodium | Cyclosporine + Mycophenolate Sodium
Started | 155 ("Started" indicates enrolled participants. Randomized participants for two arms are 154 and 146.) | 145
Completed | 118 | 117
Not Completed | 37 | 28
Not completed — Adverse Event | 19 | 9
Not completed — Lack of Efficacy | 5 | 4
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Lost to Follow-up | 0 | 8
Not completed — Administrative problems | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + Mycophenolate Sodium | Cyclosporine + Mycophenolate Sodium | Total
Number analyzed (Participants) | 155 | 145 | 300
Age Continuous [Mean (Standard Deviation); unit: Years] | 46.9 (11.67) | 46.7 (11.85) | 46.8 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 59 | 112
  Male | 102 | 86 | 188

OUTCOME MEASURES:

1. Primary Outcome: Renal Function (Nankivell Formula) at Month 12 Post Transplantation.
Description: Renal function at the end of the trial assessed as mean absolute values of the glomerular filtration rate (GFR) calculated by Nankivell formula 12 months after renal transplantation. The Nankivell formula: GFR = 6.7 / Scr + BW / 4 - Surea / 2-100 / (height)^2 + C ; where Scr is the serum creatinine concentration expressed in mmol/L, BW the body weight in kg, Surea the serum urea in mmol/L, height in m, and the constant C is 35 for male and 25 for female patients. Estimated GFR is expressed in mL/min per 1.73m^2.
Time Frame: at Month 12 post transplantation
Population: Intent to Treat Population (randomized patients); Last Observation Carried Forward (LOCF). One patient in
Measure: Mean (Standard Deviation); unit: mL/min /1.73m^2
Arm/Group | Everolimus + Mycophenolate Sodium | Cyclosporine + Mycophenolate Sodium
Number analyzed (Participants) | 154 | 145
mL/min /1.73m^2 | 71.84 (18.53) | 61.24 (16.65)

2. Secondary Outcome: Number of Participants With Occurrence of Biopsy Proven Acute Rejection (BPAR), Graft Loss or Death
Description: The number of participants with occurrence of biopsy proven acute rejection (BPAR), graft loss, or death up to Month 12 during the randomized treatment period. BPAR was defined as a biopsy graded IA, IB, IIA, IIB or III according to Banff 97 classification. A graft core biopsy was performed prior to 24 hours following initiation of graft rejection therapy. The allograft is presumed to be lost on the day the patient starts dialysis and was not able to subsequently be removed from dialysis. If the patient underwent a graft nephrectomy, then the day of nephrectomy was the day of graft loss.
Time Frame: Up to Month 12
Population: Intent to Treat Population (Randomized Patients)
Measure: Number; unit: Participants
Arm/Group | Everolimus + Mycophenolate Sodium | Cyclosporine + Mycophenolate Sodium
Number analyzed (Participants) | 154 | 146
Participants
  BPAR: Yes | 15 | 5
  BPAR: No | 139 | 141
  Graft Loss: Yes | 0 | 0
  Graft Loss: No | 154 | 146
  Death: Yes | 0 | 1
  Death: No | 154 | 145

3. Secondary Outcome: Number of Participants With Occurrence of Treatment Failures
Description: Treatment failures defined as a composite endpoint of biopsy proven acute rejection, graft loss, death, loss to follow up and discontinuations due to lack of efficacy or toxicity, or conversion to another regimen (at least one condition must be present).
Time Frame: up to or at Month 12
Population: Intention to treat (ITT) population (Randomized Patients).
Measure: Number; unit: Participants
Arm/Group | Everolimus + Mycophenolate Sodium | Cyclosporine + Mycophenolate Sodium
Number analyzed (Participants) | 154 | 146
Participants
  Treatment failure: Yes | 29 | 23
  Treatment failure: No | 125 | 123

4. Secondary Outcome: Changes in Cardiovascular Risk From Month 4.5 to Final Assessment at Month 12
Description: An updated 1991 Framingham coronary prediction algorithm was used to estimate the total risk of developing coronary heart diseases (CHD) over the course of 10 years. Risk was calculated separately for male and females. To calculate risk, points were assigned for each of the following risk factors: age, levels of LDL cholesterol, HDL cholesterol, blood pressure, cigarette smoking, and diabetes mellitus. The sum of the individual risk factor points gives a total point score, which ranges from -5 to 18 for men and -16 to 24 for women. Higher points indicate a higher risk for CHD.
Time Frame: Month 4.5 and Month 12
Population: Safety Population for whom data was available at Month 4.5 and end of treatment.
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Everolimus + Mycophenolate Sodium | Cyclosporine + Mycophenolate Sodium
Number analyzed (Participants) | 155 | 145
Points
  Male (n= 55, 37) | 0.5 (1.87) | 0.1 (1.86)
  Female (n= 22, 35) | 0.0 (2.01) | 0.8 (2.70)
  Total Population (n= 77, 72) | 0.4 (1.91) | 0.4 (2.32)

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event or Serious Adverse Event
Description: Additional information about the number of participants who experienced Adverse Events (greater than 5%) or Serious Adverse Events can be found in the Adverse Event section.
Time Frame: Aes from end of core study period (month 12) to end of follow-up period (month 60)
Population: Safety Population consisted of all participants in whom transplantation was performed and who were treated with at least one dose of any immunosuppressive medication.
Measure: Number; unit: Participants
Arm/Group | Everolimus + Mycophenolate Sodium | Cyclosporine + Mycophenolate Sodium
Number analyzed (Participants) | 155 | 145
Participants
  Adverse Events | 155 | 145
  Serious Adverse Events | 95 | 86

ADVERSE EVENTS:
Groups:
- Certican: Certican
- Sandimmun Optoral: Sandimmun Optoral
Arm/Group | Certican | Sandimmun Optoral
Serious Adverse Events (participants affected / at risk) | 103/155 | 93/145
Other Adverse Events (participants affected / at risk) | 155/155 | 145/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Certican (N=155) | Sandimmun Optoral (N=145)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 3 | 1
Myopericarditis (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 1
Amaurosis fugax (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Enteritis (Gastrointestinal disorders) | 2 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0
Peritoneal fibrosis (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Catheter site haematoma (General disorders) | 0 | 1
Fat necrosis (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 2
Hernia obstructive (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 2
Pyrexia (General disorders) | 5 | 1
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 0 | 1
Aspergilloma (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 6 | 5
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 7 | 4
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 1
Herpes zoster (Infections and infestations) | 0 | 3
Human polyomavirus infection (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 8 | 16
Pyelonephritis (Infections and infestations) | 4 | 3
Renal cyst infection (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Shunt infection (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 2 | 0
Superinfection (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 18 | 14
Urosepsis (Infections and infestations) | 5 | 4
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 2 | 0
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 3 | 7
Fat embolism (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1
Renal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Renal lymphocele (Injury, poisoning and procedural complications) | 2 | 0
Seroma (Injury, poisoning and procedural complications) | 3 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 1 | 1
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 4
Blood creatinine increased (Investigations) | 10 | 15
Blood urea increased (Investigations) | 1 | 0
Cytomegalovirus test (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Occult blood positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Tetany (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy steroid (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Dysphoria (Psychiatric disorders) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 3 | 0
IgA nephropathy (Renal and urinary disorders) | 1 | 0
Nephritis autoimmune (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Nephrosclerosis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 3 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal tubular disorder (Renal and urinary disorders) | 1 | 0
Ureteral necrosis (Renal and urinary disorders) | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 3 | 3
Urethral discharge (Renal and urinary disorders) | 1 | 0
Urethral perforation (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 2
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Urinoma (Renal and urinary disorders) | 2 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Pelvic congestion (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Kidney anastomosis (Surgical and medical procedures) | 0 | 1
Arterial restenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 3 | 2
Haemorrhage (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 9 | 14
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Certican (N=155) | Sandimmun Optoral (N=145)
Anaemia (Blood and lymphatic system disorders) | 43 | 35
Leukocytosis (Blood and lymphatic system disorders) | 17 | 22
Leukopenia (Blood and lymphatic system disorders) | 24 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 5
Vertigo (Ear and labyrinth disorders) | 7 | 9
Abdominal pain (Gastrointestinal disorders) | 20 | 14
Abdominal pain upper (Gastrointestinal disorders) | 12 | 12
Aphthous stomatitis (Gastrointestinal disorders) | 22 | 3
Constipation (Gastrointestinal disorders) | 82 | 72
Diarrhoea (Gastrointestinal disorders) | 60 | 42
Dyspepsia (Gastrointestinal disorders) | 15 | 11
Flatulence (Gastrointestinal disorders) | 25 | 20
Nausea (Gastrointestinal disorders) | 64 | 59
Vomiting (Gastrointestinal disorders) | 38 | 32
Asthenia (General disorders) | 2 | 9
Fatigue (General disorders) | 7 | 10
Impaired healing (General disorders) | 8 | 5
Oedema (General disorders) | 44 | 34
Oedema peripheral (General disorders) | 38 | 32
Pain (General disorders) | 30 | 26
Pyrexia (General disorders) | 24 | 22
Bronchitis (Infections and infestations) | 16 | 7
Cytomegalovirus infection (Infections and infestations) | 26 | 24
Gastroenteritis (Infections and infestations) | 15 | 17
Gastrointestinal infection (Infections and infestations) | 10 | 7
Herpes zoster (Infections and infestations) | 8 | 10
Human polyomavirus infection (Infections and infestations) | 8 | 3
Infection (Infections and infestations) | 9 | 9
Nasopharyngitis (Infections and infestations) | 49 | 44
Oral herpes (Infections and infestations) | 11 | 1
Pneumonia (Infections and infestations) | 16 | 9
Respiratory tract infection (Infections and infestations) | 12 | 12
Rhinitis (Infections and infestations) | 12 | 8
Upper respiratory tract infection (Infections and infestations) | 12 | 7
Urinary tract infection (Infections and infestations) | 90 | 83
Wound infection (Infections and infestations) | 4 | 11
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 21 | 24
Procedural pain (Injury, poisoning and procedural complications) | 50 | 48
Wound complication (Injury, poisoning and procedural complications) | 51 | 46
Wound dehiscence (Injury, poisoning and procedural complications) | 6 | 8
Blood creatinine increased (Investigations) | 51 | 49
C-reactive protein increased (Investigations) | 7 | 8
Weight increased (Investigations) | 8 | 14
Diabetes mellitus (Metabolism and nutrition disorders) | 19 | 12
Fluid retention (Metabolism and nutrition disorders) | 6 | 12
Hypercalcaemia (Metabolism and nutrition disorders) | 15 | 25
Hypercholesterolaemia (Metabolism and nutrition disorders) | 45 | 41
Hyperglycaemia (Metabolism and nutrition disorders) | 24 | 16
Hyperkalaemia (Metabolism and nutrition disorders) | 18 | 21
Hyperlipidaemia (Metabolism and nutrition disorders) | 23 | 16
Hyperphosphataemia (Metabolism and nutrition disorders) | 11 | 12
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 11 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 10 | 20
Hypocalcaemia (Metabolism and nutrition disorders) | 23 | 27
Hypokalaemia (Metabolism and nutrition disorders) | 45 | 36
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 47 | 43
Hypoproteinaemia (Metabolism and nutrition disorders) | 8 | 11
Iron deficiency (Metabolism and nutrition disorders) | 3 | 8
Metabolic acidosis (Metabolism and nutrition disorders) | 15 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 5
Headache (Nervous system disorders) | 25 | 21
Tremor (Nervous system disorders) | 10 | 9
Insomnia (Psychiatric disorders) | 35 | 32
Sleep disorder (Psychiatric disorders) | 21 | 20
Bladder pain (Renal and urinary disorders) | 8 | 11
Dysuria (Renal and urinary disorders) | 7 | 9
Haematuria (Renal and urinary disorders) | 28 | 31
Leukocyturia (Renal and urinary disorders) | 22 | 18
Polyuria (Renal and urinary disorders) | 10 | 16
Proteinuria (Renal and urinary disorders) | 25 | 25
Urinary retention (Renal and urinary disorders) | 11 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 17
Acne (Skin and subcutaneous tissue disorders) | 14 | 11
Hypertrichosis (Skin and subcutaneous tissue disorders) | 5 | 8
Rash (Skin and subcutaneous tissue disorders) | 8 | 4
Haematoma (Vascular disorders) | 8 | 8
Hypertension (Vascular disorders) | 17 | 22
Hypotension (Vascular disorders) | 22 | 32
Lymphocele (Vascular disorders) | 17 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.